CLINICAL TRIAL: NCT00323713
Title: Effects of Very Low Protein Diet Supplemented With Ketoanalogs on Renal Death in Phase 4/5 Chronic Kidney Disease (CKD) - ERIKA Study
Brief Title: Very Low Protein Diet and Renal Death in Chronic Kidney Disease (CKD)-ERIKA Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Sanitaria ASL Avellino 2 (Other)
Responsible Party: Dr Vincenzo Bellizzi, ASL_AV 2 - Avellino - Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA1-1425
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Renal Insufficiency
Keywords: Chronic renal insufficiency; CKD stage 4; CKD stage 5; Protein intake; Low protein diet; Very low protein diet; Ketoanalogs; Renal death
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VLPD diet (Experimental): Adavnced CKD patients (stage 4-5) on a very low protein diet
  Interventions: Behavioral: Very low protein diet
- LPD diet (Active Comparator): Adavnced CKD patients (stage 4-5) on a low protein diet
  Interventions: Behavioral: Low protein diet

INTERVENTIONS:
Behavioral: Very low protein diet — 0.3 g of proteins per kilo of body weight per day, supplemented with a mixture of essential aminoacids and chetoacids
  Other Names: VLPD
  Arms: VLPD diet
Behavioral: Low protein diet — 0.6 g of protein per kilo of body weight per day
  Other Names: LPD
  Arms: LPD diet

SUMMARY:
The purpose of this study is to determine whether the use of a very low protein diet is effective in delaying the start of chronic dialysis treatment in patients affected by chronic kidney disease (CKD).

DETAILED DESCRIPTION:
The prevalence of chronic dialysis patients is increasing worldwide because of the rising incidence of end stage renal disease, it is burdened by high cardiovascular risk, it is associated with a very high morbidity and mortality and it determines enormous costs for the community.

The improvement in the management of metabolic and cardiovascular complication associated to chronic kidney disease (CKD) since the early stages of the disease becomes mandatory in order to delay the start of dialysis and to ameliorate the whole patient outcome.

Dietary protein restriction represents a basic therapeutic approach in CKD, by reducing the accumulation of nitrogen catabolic substances, the phosphorus retention and the consequent hyperparathyroidism, the metabolic acidosis, the salt intake and the consequent hypertension, the proteinuria, and by improving the anemia and the glycemic tolerance, but the effects of the low protein diet on renal failure progression rate have not been definitely demonstrated.

Dietary effective reduction of just 0.2 g/kg/day of proteins is effective in ameliorating blood urea nitrogen, metabolic acidosis and hyperphosphoremia, and the very low protein diet (VLPD) allows a further improving of the metabolic control of uremia, it is safe, not affecting the nutritional status, and it is cost saving. VLPD has been suggested to delay the start of renal replacement therapy with respect to standard low protein diet, by mean of either secondary analysis of clinical trials or retrospective analysis.

Large randomized clinical trials (RCT) on this issue lack, and the effect of VLPD on renal death remain to be addressed. As well, information on patients' compliance to VLPD prescription and on the impact of VLPD on the quality of life are needed. Finally, also the effects of VLPD on both cardiovascular risk factors and mortality remain to be completely evaluated.

The primary aim of this study is to evaluate, by mean of a RCT, the effect of the very low protein diet on the renal death in renal patients affected by chronic renal insufficiency of moderate to advanced degree (CKD stages 4 and 5). Secondary aims are to evaluate the effect of VLPD on cardiovascular risk factors, morbidity and mortality, the adherence to VLPD, and the relationship between VLPD and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal insufficiency in stage CKD 4 and 5 (GFR < 30 ml/min/1.73m2, estimated by the 24-hours creatinine clearance) receiving conservative treatment for CKD
* Incident patients with chronic renal insufficiency in stage CKD 4 and 5 (GFR < 30 ml/min/1.73m2, estimated by the 24-hours creatinine clearance), provided stable renal function determined by two 24-hour measurements of creatinine clearance 2 weeks a part

Exclusion Criteria:

* Patients already on very low protein diet
* Change of creatinine clearance > 30% within the last 3 months
* Severe undernutrition as indicated by :

  1. BMI < 20 kg/m2 in presence of serum albumin < 3.0 g/dl, or BMI < 17.5 kg/m2 whatever albumin value
  2. body weight reduction > 7.5% within the last 3 months
* Severe obesity as indicated by BMI > 35 kg/m2
* Pregnancy or feeding
* Chronic treatment with steroid or cytotoxic drugs
* Fast progressing glomerulonephritis
* Active SLE and vasculitis
* Cardiac failure stage IV NYHA
* Advanced liver cirrhosis
* Active cancer diseases
* Severe encephalopathy associated with lack of spontaneous feeding
* Chronic obstructive respiratory diseases needing oxygen treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2005-02; Primary Completion 2011-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Time to renal death, defined as the first event between start of renal replacement therapy or patient death | Months

SECONDARY OUTCOMES:
Compliance to diet | Months
Quality of life | Months
Cardiovascular morbidity, defined by angina, heart failure, myocardial infarction, left ventricular mass, stroke, blood pressure, lipid profile, calcium/phosphorus/parathormone status and Charlson comorbidity index, at the start of dialysis | Months
Nutritional status, defined by anthropo-plicometry, biochemistry, body bioimpedance analysis (BIA), subjective global nutritional assessment (SGA), at the start and during the 1st year of dialysis | Months
Cardiovascular mortality | Months

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Bellizzi, MD, PhD, Study Chair — Nephrology Unit "A. Landolfi" Hospital, Solofra (AV) Italy; Giuseppe Conte, MD, Study Chair — Division of Nephrology, Medical School, Second University of Naples, Naples, Italy; Ciro Gallo, MD, Study Chair — Biostatistics Unit, Medical School, Second University of Naples, Naples, Italy
Locations (17):
- Italy (17):
  - Nephrology Unit, "Moscati" Hospital, Avellino, AV
  - Nephrology Unit, S. Angelo dei Lombardi Hospital, Sant'Angelo dei Lombardi, AV
  - Nephrology Unit "A. Landolfi" Hospital, Solofra, AV
  - Nephrology Division, Medical School, University of Bari, Bari, BA
  - Nephrology Unit, Brindisi Hospital, Brindisi, BR
  - Nephrology Unit, Piedimonte Matese Hospital, Piedimonte Matese, CE
  - Nephrology Unit, S. Felice a Cancello Hospital, San Felice A Cancello, CE
  - Nephrology Division, Medical School, University of Catanzaro, Catanzaro, CZ
  - Nephrology Division, Medical School, University of Foggia, Foggia, FG
  - Nephrology Unit, Foggia Hospital, Foggia, FG
  - Nephrology Unit, San Severo Hospital, San Severo, FG
  - Nephrology Unit, Galatina Hospital, Galatina, LE
  - Nephrology Division, "San Carlo" Hospital, Potenza, PZ
  - Nephrology Unit, "Curto" Hospital, Polla, SA
  - Nephrology Unit, Castellammare Hospital, Castellammare di Stabia
  - Nephrology Division, Medical School, University "Federico II" of Naples, Napoli
  - Nephrology Division, Medical School, Second University of Naples, Napoli

REFERENCES:
- [Background] Di Iorio BR, Minutolo R, De Nicola L, Bellizzi V, Catapano F, Iodice C, Rubino R, Conte G. Supplemented very low protein diet ameliorates responsiveness to erythropoietin in chronic renal failure. Kidney Int. 2003 Nov;64(5):1822-8. doi: 10.1046/j.1523-1755.2003.00282.x. PMID 14531817
- [Background] Di Iorio BR, Bellizzi V, Minutolo R, De Nicola L, Iodice C, Conte G. Supplemented very low-protein diet in advanced CRF: is it money saving? Kidney Int. 2004 Feb;65(2):742. doi: 10.1111/j.1523-1755.2004.404_2.x. No abstract available. PMID 14717953
- [Background] Bellizzi V, Di Iorio BR, De Nicola L, Minutolo R, Zamboli P, Trucillo P, Catapano F, Cristofano C, Scalfi L, Conte G; ERIKA Study-group. Very low protein diet supplemented with ketoanalogs improves blood pressure control in chronic kidney disease. Kidney Int. 2007 Feb;71(3):245-51. doi: 10.1038/sj.ki.5001955. Epub 2006 Oct 11. PMID 17035939
- [Derived] Hahn D, Hodson EM, Fouque D. Low protein diets for non-diabetic adults with chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 29;10(10):CD001892. doi: 10.1002/14651858.CD001892.pub5. PMID 33118160